CLINICAL TRIAL: NCT03045874
Title: Community Partnership for Healthy Sleep
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1510016673; R21NR016190-01A1 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-08 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Pediatric Sleep

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 30 parent-child dyads: Stratified purposive sampling will assure representation proportional to the minority representation in the community and will include equal subsamples (15 families each) of families with children 6-18 months of age and children aged 19-36 months.
- 30 primary care providers: Investigators will purposively recruit 30 primary care providers to assure proportional representation of physicians and NPs with a "snowball" method. The sample sizes should be sufficient to achieve saturation of the data for qualitative analyses, but we will recruit more participants if saturation is not obtained with the planned sample.
- focus groups: The investigators will hold separate focus groups for parents of the two age groups and clinicians. We anticipate conducting approximately 6 focus groups with 8-10 participants in each to review and refine the sleep program.
- 22 parent-child dyads: The investigators will conduct feasibility testing of a 3 week sleep health promotion intervention. The intervention will be delivered to parents of children ages 12-36 months enrolled in one childcare center.
- 5 childcare teachers: Teachers will be trained to deliver a brief sleep health intervention

SUMMARY:
The purpose of this study is to conduct community-engaged research (CEnR) with families and pediatric providers caring for the children in those families to address the following specific aims:

1. Examine parents' knowledge and perceptions about their 6-36 month old children's sleep and objective characteristics of sleep, including (1a) self-reported and actigraph-recorded characteristics of sleep, sleep habits, and difficulty; (1b) the contributions of sleep habits and individual, family, community, cultural/social, and health-related factors to sleep characteristics and sleep difficulty; (1c) consequences of sleep difficulty; (1d) successful and unsuccessful strategies used to promote children's sleep and sleep habits; (1e) preferences regarding sleep promotion interventions for their children; and perceptions of the optimal timing to begin sleep promotion intervention
2. Examine pediatric primary care providers' perceptions about (2a) the importance of sleep and sleep habits for 6-36 month old children; (2b) factors that contribute to sleep habits and sleep difficulty; (2c) successful and unsuccessful approaches to promote healthy sleep habits, adequate duration and good quality sleep and assessment and management of sleep difficulty in young children within the context of their families; and (2c) barriers, facilitators, and preferences regarding sleep-promoting interventions for families with young children;
3. Collaborate with families and providers to use the information obtained in Aims 1 and 2 to develop and refine a feasible, relevant, and acceptable sleep promotion program, including procedures, protocols, patient materials, intervention fidelity plans, and delivery methods.

DETAILED DESCRIPTION:
The investigators will conduct this study in 3 phases, employ Community Engaged Research (CEnR), and use guidelines for community participation developed through Yale Center for Clinical Investigation (YCCI/Yale's CTSA). The Social Ecological Model, depicting interactions among the environment, individual, family, community, and society as they influence health, will guide the study. The key informants and community and clinical stakeholders represent layers of the model49-51 acknowledging the critical intersection between the model components and health promotion behavior (i.e., healthy sleep habits).

Community Engagement. The investigators will extend the CEnR process begun in our preliminary work to engage two groups of community stakeholders: parents of children between the ages of 6-36 months and pediatric primary care clinicians who provide health care to those children. The investigators will invite 8-10 volunteers (pediatricians, nurse practitioners, parents of 6-18 month old children, parents of 19-36 month olds) to join our team as members of a Community Advisory Committee that will meet quarterly throughout this project to assist with oversight and share decision-making about methods, interpretation of findings, and intervention development, implementation, evaluation, and dissemination. The investigators will meet at convenient times and locations and use conference calls if preferred. The investigators will compensate parents and providers for time spent in study activities and reimburse parents for taxi cab fare. The investigators will provide onsite childcare in a separate room from the interviews. The investigators will offer committee members co-authorship on reports and collaboration on disseminating information on sleep habits into the community. The investigators will also invite them to continue to guide future studies and intervention projects. Consistent with a CEnR approach, The investigators will include them as full partners in future collaborations as preferred.

In Phase I/Aims 1 & 2 the investigators will employ a convergent mixed methods approach in which the investigators will collect quantitative (questionnaires) and qualitative interview data (semi-structured interview) about parents' perceptions of children's sleep, sleep habits, sleep difficulty, and sleep-promoting interventions (Aim 1). The investigators will also use semi-structured interviews to elicit perceptions about the importance of sleep, promotion of healthy sleep habits, sleep assessment, sleep difficulties, and barrier and facilitators to sleep promotion, assessment, and intervention from primary care clinicians (Aim 2).

In Phase II/Aim 3 the investigators will collaborate with the Community Advisory Board to draft a sleep promotion program, based on phase I results and the literature. Deliverables will include objectives, content, procedures, protocols, patient materials, intervention fidelity procedures, and delivery methods, including a possible prototype of an mHealth approach. The investigators will use an iterative method, including focus groups with our two communities, for member checking and cognitive interviewing to assess feasibility, cultural relevance and acceptability of the intervention. Investigators will conduct feasibility testing of the sleep promotion intervention in one childcare center.

ELIGIBILITY:
Inclusion Criteria for parents:

* fluent in English
* New Haven residents
* obtain pediatric care in a New Haven community practice
* parents of 6-18 month old children
* parents of 19-36 month old children

Exclusion Criteria for parents:

* severe mental illness
* severe cognition impairment
* substance-related symptoms requiring inpatient hospitalization or ambulatory detoxification
* those whose children have a serious illness, significant developmental delays
* parents with children in custody of the CT Department of Children and Family Services

Inclusion Criteria for Pediatric primary care providers

* experienced in the care of community children
* provide care in the greater New Haven are
* speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents will reside in New Haven and obtain pediatric health care in a New Haven community practice.
  Pediatric primary care providers will be experienced in the care of community children and will include physicians, senior resident pediatricians, and nurse practitioners (NPs) who provide primary care in the greater New Haven area and speak English.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
parent knowledge about sleep | interview of approximately 60 minutes
  A member of the research team experienced in qualitative interviewing will conduct the parent interviews in a private space at the PCC, Yale School of Nursing (YSN), or other convenient location at a time separate from a health care visit. Investigators will use a semi-structured guide organized by the constructs of interest (e.g. sleep characteristics, importance of sleep, sleep habits, contributing factors). Open-ended prompts will be used to explore ideas.
  Interview data will be digitally transcribed and uploaded into Atlas.ti software. Investigators will use a qualitative descriptive approach and a constant comparative method in which data collection and analysis occur simultaneously to allow for a flexible and emergent design, with modification of the interview schedule and probes as new patterns or directions emerge from the data.
parent distress/stress via Brief Symptom Inventory (BSI) | interview of approximately 60 minutes
  The 18-item BSI includes a Global Severity Index (GSI: symptomatology across multiple domains during the preceding 2 week) and subscales (depression, somatization and anxiety symptoms).
actigraph sleep duration | 9 nights
  Objective sleep characteristics will be measured with the Respironics Minimitter Actiwatch AW2. Reliability for actigraphy in 12-24 month old children ranges from .67-.85 (sleep duration) and .77-.89 (efficiency). As in earlier studies, the actigraph will be worn on the ankle. The parent will depress the event marker at "lights out"/bedtime, "lights on," and naptime and record the times in the diary. A user-friendly guide will be used to explain this process to parents. The investigators will phone parents every two days to address questions and remind them to continue. The investigators will request 9 days and nights of data to obtain at least seven nights, a period that will enable us to determine daily variability.
actigraph sleep efficiency | 9 nights
  Objective sleep characteristics will be measured with the Respironics Minimitter Actiwatch AW2. Reliability for actigraphy in 12-24 month old children ranges from .67-.85 (sleep duration) and .77-.89 (efficiency). As in earlier studies, the actigraph will be worn on the ankle. The parent will depress the event marker at "lights out"/bedtime, "lights on," and naptime and record the times in the diary. A user-friendly guide will be used to explain this process to parents. The investigators will phone parents every two days to address questions and remind them to continue. The investigators will request 9 days and nights of data to obtain at least seven nights, a period that will enable us to determine daily variability.
actigraph nap duration | 9 days
  Objective sleep characteristics will be measured with the Respironics Minimitter Actiwatch AW2. Reliability for actigraphy in 12-24 month old children ranges from .67-.85 (sleep duration) and .77-.89 (efficiency). As in earlier studies, the actigraph will be worn on the ankle. The parent will depress the event marker at "lights out"/bedtime, "lights on," and naptime and record the times in the diary. A user-friendly guide will be used to explain this process to parents. The investigators will phone parents every two days to address questions and remind them to continue. The investigators will request 9 days and nights of data to obtain at least seven nights, a period that will enable us to determine daily variability.
parent-reported sleep patterns | interview of approximately 60 minutes
  by diary and interview, Interview data will be digitally transcribed and uploaded into Atlas.ti software. Investigators will use a qualitative descriptive approach and a constant comparative method in which data collection and analysis occur simultaneously to allow for a flexible and emergent design, with modification of the interview schedule and probes as new patterns or directions emerge from the data.
parent stress/distress via Parenting Stress Index (PSI)-Short Form | interview of approximately 60 minutes
  The BSI is reliable and valid (GSI alpha = 0.90), requires a 6th grade reading level, and the investigators have used it in studies with adolescent and young parents.69 The 36 item PSI-short form, 83 a measure of the relative magnitude of stress in the parent-child system is rated on a 5 point scale and yields five subscale scores: Parent Distress, Parent-Child Difficulty, Difficult Child, Defensive Responding, and Total Stress. The PSI subscales have concurrent validity with the full-length PSI.84 Alpha coefficients ranged from.88-.95- across the five subscales in similar samples

SECONDARY OUTCOMES:
perceptions of the importance of sleep from providers | interview of approximately 60 minutes
  Interview and focus group data will be digitally transcribed and uploaded into Atlas.ti software. The investigators will use a qualitative descriptive approach and a constant comparative method in which data collection and analysis occur simultaneously to allow for a flexible and emergent design, with modification of the interview schedule and probes as new patterns or directions emerge from the data.
successful and unsuccessful approaches to promoting healthy sleep habits from providers | interview of approximately 60 minutes
  Interview and focus group data will be digitally transcribed and uploaded into Atlas.ti software. The investigators will use a qualitative descriptive approach and a constant comparative method in which data collection and analysis occur simultaneously to allow for a flexible and emergent design, with modification of the interview schedule and probes as new patterns or directions emerge from the data.
assessing and managing sleep disorders from providers | interview of approximately 60 minutes
  Interview and focus group data will be digitally transcribed and uploaded into Atlas.ti software. The investigators will use a qualitative descriptive approach and a constant comparative method in which data collection and analysis occur simultaneously to allow for a flexible and emergent design, with modification of the interview schedule and probes as new patterns or directions emerge from the data.
resources needed to support assessment and management from providers | interview of approximately 60 minutes
  Interview and focus group data will be digitally transcribed and uploaded into Atlas.ti software. The investigators will use a qualitative descriptive approach and a constant comparative method in which data collection and analysis occur simultaneously to allow for a flexible and emergent design, with modification of the interview schedule and probes as new patterns or directions emerge from the data.
barriers, facilitators, and preferences for sleep-promoting interventions from providers | interview of approximately 60 minutes
  Interview and focus group data will be digitally transcribed and uploaded into Atlas.ti software. The investigators will use a qualitative descriptive approach and a constant comparative method in which data collection and analysis occur simultaneously to allow for a flexible and emergent design, with modification of the interview schedule and probes as new patterns or directions emerge from the data.
focus group to assess feasibility, cultural relevance and acceptability | 90 minutes
  Investigators will hold separate focus groups for parents of the two age groups and clinicians. The investigators anticipate conducting approximately 6 focus groups with 8-10 participants in each to review and refine the sleep program.
  The investigators will use an iterative method, including focus groups with our two communities, for member checking and cognitive interviewing, to assess feasibility, cultural relevance and acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Redeker, PhD, Principal Investigator — Yale School of Nursing; Lois Sadler, PhD, Principal Investigator — Yale School of Nursing
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ordway MR, Sadler LS, Jeon S, O'Connell M, Banasiak N, Fenick AM, Crowley AA, Canapari C, Redeker NS. Sleep health in young children living with socioeconomic adversity. Res Nurs Health. 2020 Aug;43(4):329-340. doi: 10.1002/nur.22023. Epub 2020 Apr 19. PMID 32306413